CLINICAL TRIAL: NCT03495817
Title: An Open-Label Safety, Tolerability, and Efficacy Study in Male and Female Subjects With Androgenetic Alopecia Treated With ATI-50002 Topical Solution
Brief Title: A Study in Male and Female Subjects With Androgenetic Alopecia Treated With ATI-50002 Topical Solution
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-50002-AGA-201
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ATI-50002 Topical Solution (Experimental): This is an open-label phase 2 study designed to evaluate the safety and efficacy of ATI- 50002 Topical Solution, 0.46% in male and female subjects with androgenetic alopecia.
  Subjects will be required to apply ATI-50002 study medication to their scalp twice a day for a total of 26 weeks.
  Interventions: Drug: ATI-50002

INTERVENTIONS:
Drug: ATI-50002 — ATI-50002 Topical Solution

SUMMARY:
Open label study to assess safety, tolerability, and efficacy of ATI-50002 in male and female subjects with androgenetic alopecia.

DETAILED DESCRIPTION:
This is an open-label study designed to evaluate the safety and efficacy of ATI-50002 Topical Solution in male and female subjects with androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

Male subjects and non-pregnant, non-nursing female subjects 18-50 years of age with a clinical diagnosis of androgenetic alopecia.

Subjects willing to agree to have a small circle of hair clipped to approx. 1mm in length on their balding spot.

Subjects willing to agree to have a permanent dot tattoo applied to their scalp to mark the center of the identified target area.

Subjects must agree to maintain the same hair style and hair care regimen during the study.

Exclusion Criteria:

Females who are nursing, pregnant, or planning to become pregnant for the duration of the study and up to 30 days after the last application of study medication.

Clinical diagnosis of alopecia areata or other non AGA forms of alopecia. Scalp hair loss on the treatment area, due to disease, injury or medical therapy.

Active skin disease of the scalp (such as psoriasis or seborrheic dermatitis) or a history of skin disease on the scalp that in the opinion of the investigator would interfere with the study assessments or efficacy or safety.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Shanler, MD, Study Chair — Aclaris Therapeutics, Inc.
Locations (3):
- United States (3):
  - Aclaris Investigational Site, Denver, Colorado
  - Aclaris Investigational Site, Portland, Oregon
  - Aclaris Investigational Site, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- ATI-50002 Topical Solution: This is an open-label phase 2 study designed to evaluate the safety and efficacy of ATI-50002 Topical Solution, 0.46% in male and female subjects with androgenetic alopecia.
  Upon completion of the first 26 weeks of treatment, subjects will have the option to consent to continue on study medication for an additional 26 weeks of treatment.
  Subjects will be required to apply ATI-50002 study medication to their scalp twice a day for a total of 26 weeks.
Period: 26 Week Open Label
Arm/Group | ATI-50002 Topical Solution
Started | 31
Completed | 23
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Period: 26 Week Extension
Arm/Group | ATI-50002 Topical Solution
Started (The 26-week extension was not required, and 4 patients elected to not start the extension.) | 19
Completed | 17
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (6.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity was only self-reported for those participants identifying as "White".
  Participants
    number analyzed (Participants) | 25
    Hispanic or Latino | 3
    Not Hispanic or Latino | 21
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 1
  White | 25
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 31
Height [Mean (Standard Deviation); unit: centimeters] | 173.7 (9.04)
Weight [Mean (Standard Deviation); unit: kilograms] | 89.4 (20.74)
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - Always Burns | 3
  II - Burns Easily | 11
  III - Burns Moderately | 10
  IV - Burns Minimally | 4
  V - Rarely Burns | 2
  VI - Never Burns | 1
Sinclair Grade (Females) [Count of Participants; unit: Participants] — Treating investigators will be required to rate the subject's level of hair loss at baseline based on the Sinclair scale for women.
  Grade 1: is normal. This pattern is found in all girls prior to puberty but in only forty-five percent of women aged eighty or over.
  Grade 2: shows a widening of the central part. Grade 3: shows a widening of the central part and thinning of the hair on either side of the central part.
  Grade 4: reveals the emergence of a diffuse hair loss over the top of the scalp.
  Grade 5: indicates advanced hair loss. Population: Sinclair grading only applies to those participants that are Female.
  Participants
    number analyzed (Participants) | 10
    Grade 1 | 0
    Grade 2 | 4
    Grade 3 | 4
    Grade 4 | 2
    Grade 5 | 0
Norwood-Hamilton Classification [Count of Participants; unit: Participants] — Subject's level of hair loss at baseline based on the Norwood Hamilton Scale for male subjects.
  Type I: Minimal or no recession of the hairline Type II: Triangular areas of recession at the frontotemporal hairline Type III: Deep symmetrical recession at the temples are bare or only sparsely covered by hair Type IV: Frontotemporal recession is more severe than in Type III with sparse or no hair on the vertex Type V: The vertex hair loss region is separated from the frontotemporal region but is less distinct Type VI: Sparse hair remaining Type VII: The most severe form of hair loss Population: Norwood-Hamilton Classification only applies to those participants that are Male.
  Participants
    number analyzed (Participants) | 21
    Type I | 0
    Type II | 0
    Type III | 7
    Type IV | 5
    Type V | 9
    Type VI | 0
    Type VII | 0
Prior Therapies for Androgenetic Alopecia [Count of Participants; unit: Participants] — A single study patient may have tried more than one prior therapy.
  Participants
    Device | 2
    Finasteride | 2
    Investigational Medication (Oral) | 1
    Investigational Medication (Topical) | 1
    Minoxidil | 4
    Other | 7
    No Prior Therapy | 20
Time since Diagnosis of Androgenetic Alopecia [Mean (Standard Deviation); unit: years] | 7.89 (5.098)
Age at Diagnosis of Androgenetic Alopecia [Mean (Standard Deviation); unit: years] | 30.4 (8.05)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Target Area Hair Count (TAHC)
Description: Target Area Hair Count will measure the hairs/cm2 on a subject's head. Higher values represent better outcomes.
Time Frame: Baseline to 26 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Mean (Standard Deviation); unit: hairs/cm^2
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 20
hairs/cm^2 | 8.6 (12.87)

2. Secondary Outcome: Mean Change From Baseline in Target Area Hair Count (TAHC)
Description: Target Area Hair Count will measure the hairs/cm2 on a subject's head. Higher values represent better outcomes.
Time Frame: Baseline to 52 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Mean (Standard Deviation); unit: hairs/cm^2
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 17
hairs/cm^2 | 1.6 (18.92)

3. Secondary Outcome: Mean Change From Baseline in Cumulative Target Area Hair Width (TAHW)
Description: Target Area Hair Width (TAHW) will measure the cumulative width of hair in the subject's target area. Higher values represent better outcomes.
Time Frame: Baseline to 26 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 20
microns | 403.69 (817.271)

4. Secondary Outcome: Mean Change From Baseline in Cumulative Target Area Hair Width (TAHW)
Description: as for outcome 3
Time Frame: Baseline to 52 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 17
microns | 35.28 (901.082)

5. Secondary Outcome: Investigator Global Assessment: Total Subjects With Slightly Increased Hair Growth or Better Using a Seven-point Rating Scale
Description: Investigators will use a 7 point rating scale to assess hair growth following treatment with study medication. A score of +3 corresponds to significant hair growth and a score of -3 corresponds to lack of hair growth. Subjects with a score of +1 to +3 were considered to have slightly increased hair growth or better.
Time Frame: Baseline to 26 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 22
Participants | 16

6. Secondary Outcome: Investigator Global Assessment: Total Subjects With Slightly Increased Hair Growth or Better Using a Seven-point Rating Scale
Description: as for outcome 5
Time Frame: Baseline to 52 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 12
Participants | 8

7. Secondary Outcome: Subject Self-Assessment: Total Subjects With Slightly Increased Hair Growth or Better Using a Seven-point Rating Scale
Description: Subjects will use a 7 point rating scale to assess hair growth following treatment with study medication. A score of +3 corresponds to significant hair growth and a score of -3 corresponds to lack of hair growth. Subjects with a score of +1 to +3 were considered to have slightly increased hair growth or better.
Time Frame: Baseline to 26 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 22
Participants | 18

8. Secondary Outcome: Subject Self-Assessment: Total Subjects With Slightly Increased Hair Growth or Better Using a Seven-point Rating Scale
Description: as for outcome 7
Time Frame: Baseline to 52 Weeks
Population: The variation in total number of patients reported across the various assessments is due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 17
Participants | 13

9. Secondary Outcome: Change From Baseline in Androgenetic Alopecia (AGA) Using the Norwood-Hamilton Scale
Description: Measure Description: Subject's level of hair loss at baseline based on the Norwood Hamilton Scale for male subjects.
  Type I: Minimal or no recession of the hairline Type II: Triangular areas of recession at the frontotemporal hairline Type III: Deep symmetrical recession at the temples are bare or only sparsely covered by hair Type IV: Frontotemporal recession is more severe than in Type III with sparse or no hair on the vertex Type V: The vertex hair loss region is separated from the frontotemporal region but is less distinct Type VI: Sparse hair remaining Type VII: The most severe form of hair loss. Lower scores represent better outcomes.
Time Frame: Baseline to 26 Weeks
Population: This measurement only applies to men participating in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 15
Participants
  Improvement from Type V to Type III Vertex | 2
  Improvement from Type V to Type IV | 1
  Improvement from Type IV to Type III Vertex | 1
  Improvement from Type III to Type III Vertex | 2
  No Improvement Measured | 9

10. Secondary Outcome: Change From Baseline in Androgenetic Alopecia (AGA) Using the Norwood-Hamilton Scale
Description: as for outcome 9
Time Frame: Baseline to 52 Weeks
Population: This measurement only applies to men participating in the study. Variances from participant low section are the result of missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 14
Participants
  Improvement from Type V to Type III Vertex | 1
  Improvement from Type III Vertex to Type II | 1
  Improvement from Type V to Type IV | 1
  Improvement from Type IV to Type III Vertex | 1
  Improvement from Type III Vertex to Type III | 1
  No Improvement | 9

11. Secondary Outcome: Change From Baseline in Androgenetic Alopecia (AGA) Using the Sinclair Scale
Description: Treating investigators will be required to rate the subject's level of hair loss at baseline based on the Sinclair scale for women.
  Grade 1: is normal. This pattern is found in all girls prior to puberty but in only forty-five percent of women aged eighty or over.
  Grade 2: shows a widening of the central part. Grade 3: shows a widening of the central part and thinning of the hair on either side of the central part.
  Grade 4: reveals the emergence of a diffuse hair loss over the top of the scalp.
  Grade 5: indicates advanced hair loss. Lower grades represent better outcomes.
Time Frame: Baseline to 26 Weeks
Population: This measurement only applies to women participating in the study. Variances from participant low section are the result of missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 7
Participants
  Improvement from Grade 4 to Grade 3 | 1
  Improvement from Grade 2 to Grade 1 | 1
  No Measured Improvement | 5

12. Secondary Outcome: Change From Baseline in Androgenetic Alopecia (AGA) Using the Sinclair Scale
Description: as for outcome 11
Time Frame: Baseline to 52 Weeks
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | ATI-50002 Topical Solution
Number analyzed (Participants) | 3
Participants
  Improvement from Grade 4 to Grade 3 | 1
  Improvement from Grade 3 to Grade 2 | 1
  No Improvement | 1

ADVERSE EVENTS:
Time Frame: Open Label = 26 weeks; Extension period = 26 weeks; Reporting of non-serious AEs started with each subject's first study medication application and continued until 30 days following the last application of study medication. Events with onset dates more than 30 days after the last application of study medication were considered as "post-therapy."
Arm/Group | ATI-50002 Topical Solution
All-Cause Mortality (participants affected / at risk) | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 18/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-50002 Topical Solution (N=31)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ATI-50002 Topical Solution (N=31)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Photopsia (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Nasal herpes (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT03495817/Prot_000.pdf
  • Informed Consent Form (2018-10-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03495817/ICF_001.pdf
  • Statistical Analysis Plan (2019-04-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT03495817/SAP_002.pdf